CLINICAL TRIAL: NCT01317017
Title: Cellular Responses To Intradermal-Gamma (IFN-gamma) in Normal and Psoriatic Patients
Brief Title: Cell Responses to IFN-gamma
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Unable to isolate sufficient cells from the skin biopsy to perform study experiments.
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MLO-0717
Record Dates: First submitted 2011-03-10; First posted 2011-03-16 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — interferon gamma-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Actimmune — * All subjects will receive one intradermal injections of 0.25ml of IFN-g (Actimmune TM 100 micrograms/0.5ml), in normal appearing skin of both normal volunteers and psoriasis patients.
  * Blood will be taken at baseline and day 1. A skin biopsy (6mm punch) will be taken at the injection site 24 hours later.
  * Patients will return at one to two weeks for suture removal.
  * Clinical assessments done at every visit.
  * Patients will also be evaluated at each visit for any adverse events.

SUMMARY:
IFN-gamma is a central player in the development of psoriasis lesions, which can be involved a variety of cellular processes in the skin. Dendritic cells are important cells in driving inflammation in psoriasis through the induction of T cells that produce IL-17 in psoriasis. Injecting IFN-g into the skin can increase the numbers of T cells and also inflammatory DCs that produce cytokines involved in IL-17 production. Thus, the investigators hypothesize that the dendritic cells present in the skin after IFN-g injection polarize IL-17-producing T cells.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Normal volunteers with no evidence of skin disease OR diagnosis of plaque type psoriasis for at least 6 months
* 18 years of age or greater
* For women of childbearing potential or in men whose partners may become pregnant, willingness to use an acceptable method of contraception to prevent pregnancy for the duration of the study. Acceptable methods of contraception include use of a condom; abstinence; use by sexual partner of oral implantable or injectable contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap; or a sterile sexual partner

Exclusion Criteria:

* Guttate, erythrodermic, or pustular psoriasis as sole or predominant form of psoriasis
* Clinically significant psoriasis flare during screening or on the first treatment day
* Hypersensitivity to IFN-g or E. coli derivatives
* Pre-existing, uncontrolled myelosuppression, cardiac disease, seizure disorders, compromised central nervous system function or multiple sclerosis
* History of malignancy, clinically significant renal insufficiency, poorly controlled medical conditions that would increase the risks
* Presence of malignancy within the past 5 years, including lymphoproliferative disorders. Subjects with a history of fully resolved basal cell or squamous cell skin cancer may be enrolled.
* Pregnancy or lactation. As the risk of IFN-g in pregnancy is unknown, pregnant women will be excluded from the study.
* Any medical condition that, in the judgment of the investigator, would jeopardize the subject's safety following exposure to study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Function of dendritic cells from IFNg-injected skin | 6 months
  To perform an assay using dendritic cells from the biopsy as stimulator cells and T cells as responders.

SECONDARY OUTCOMES:
Flow cytometry analysis of circulating leukocyte populations | 9 months
  Surface phenotype and intracellular cytokine staining will be performed to determine if a single dose of IFNg alters circulating leukocyte phenotype.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Lowes, MD, Principal Investigator — The Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States